CLINICAL TRIAL: NCT04156425
Title: The Role of PKC Activation in the Immune-inflammatory Mechanism of Major Depressive Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 81930033
Record Dates: First submitted 2019-10-29; First posted 2019-11-07 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-10

CONDITIONS: Major Depressive Disorder
Keywords: Major Depressive Disorder; neuroimmunology; Protein Kinase C
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: group1：escitalopram + golimumab (N = 60), group2：escitalopram + calcium tablet (N = 60) group3：escitalopram +placebo (N = 60).
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- escitalopram + golimumab (Experimental): Patients will be treated with escitalopram from the minimum dosage and golimumab according to direction for use.
  Interventions: Drug: Escitalopram+golimumab
- escitalopram + calcium tablet (Experimental): Patients will be treated with escitalopram from the minimum dosage and calcium tablet according to direction for use.
  Interventions: Dietary Supplement: Escitalopram+Calcium Tablet
- escitalopram (Active Comparator): Patients will be treated with escitalopram from the minimum dosage.
  Interventions: Drug: Escitalopram

INTERVENTIONS:
Drug: Escitalopram+golimumab — Escitalopram will be administered at 10-20 mg/d during the acute phase. Golimumab will be administered at the dose of 50mg every month during the acute phase.
  Other Names: Lexapro+Simponi
  Arms: escitalopram + golimumab
Dietary Supplement: Escitalopram+Calcium Tablet — Escitalopram will be administered at 10-20 mg/d during the acute phase. Calcium tablet will be administered at 2000mg/d during the acute phase.
  Other Names: Lexapro+Caltrate
  Arms: escitalopram + calcium tablet
Drug: Escitalopram — Escitalopram will be administered at 10-20 mg/d during the acute phase.
  Other Names: Lexapro
  Arms: escitalopram

SUMMARY:
Major Depressive disorder (MDD) is a heterogeneous mental illness. Treated with antidepressants that act on the neurotransmitter and/or their receptors just remitted only one third of patients with MDD, Thus, to improve the efficacy is a major unmet need for depression. Based on the scientific reports, inflammation plays a definite role in the development and treatment of depression, which may be an important way to understand and finally solve the problem. Our team found that there were significant changes in tumor necrosis factor (TNF)-α and other inflammatory factors in depressed patients, which caused neuronal apoptosis and depressive symptoms; PRKCB1(gene of protein kinase C-β) plays an anti-inflammatory role by regulating protein kinase C(PKC) activation in specific brain region, improving neuroplasticity and playing an antidepressant role. In this study, we assumes that the treatment-resistant depression patients maybe due to the immune inflammation and PKC activation inconsistency or unsynchronized, which couldn't reversible microglia polarization and neuronal apoptosis in specific brain regions, then, caused the significant changes at emotional and cognitive neural circuits, so as to exhibit such as emotional, cognitive symptoms of depression. Therefore, activating PKC and regulating immune/inflammatory process will be another way to improve the treatment outcome of depression. Take consideration, we focus on treatment-resistant depression patients, to validate the relationship between PKC activation and the immune inflammatory mechanism of depression, evaluate the antidepressant effect of golimumab or calcium tablet (a PKC activator) plus escitalopram, and initially proposes idividualized treatment strategies for MDD.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled antidepressant augmentation trial. All participants are randomly divided into 3 groups treated orally with "escitalopram + golimumab" (N = 60), "escitalopram + calcium tablet" (N = 60) or "escitalopram +placebo" (N = 60).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men or women of matched age, gender and education with that of treatment-resistant depression (TRD) group;
2. A willingness to adhere to all prohibitions and restrictions necessary for the study;
3. Signed informed consent.

Exclusion Criteria:

1. Participant who have severe mental diseases, physical diseases, cerebrovascular disease, or a history of traumatic brain injury;
2. Participant who had a serious allergic reaction disease or those who have suffered from diseases of the immune system;
3. Participant who used anti-inflammatory drugs, or immunomodulatory drugs no more than 1 month prior randomization;
4. Pregnant or lactating female.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 180 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
remission of acute phase | 12th week
  scored 7 or lower on the Hamilton's Depression Scale with 17 items

CONTACTS AND LOCATIONS:
Overall Officials: Yiru Fang, Study Chair — Shanghai Mental Health Center

REFERENCES:
- [Derived] Guo X, Mao R, Cui L, Wang F, Zhou R, Wang Y, Huang J, Zhu Y, Yao Y, Zhao G, Li Z, Chen J, Wang J, Fang Y. PAID study design on the role of PKC activation in immune/inflammation-related depression: a randomised placebo-controlled trial protocol. Gen Psychiatr. 2021 Apr 5;34(2):e100440. doi: 10.1136/gpsych-2020-100440. eCollection 2021. PMID 33912799